CLINICAL TRIAL: NCT04321564
Title: Comparison of Beck Depression Score in Multipar and Nulliparous Women Who Have Gone Under Dilatation and Curettage
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.7.17
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Depression; Anxiety Depression; Pregnancy Early
Keywords: Beck Depression; Beck Anxiety; parite; curettage
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nullipar pregnant women
- multipar pregnant women

SUMMARY:
It is aimed to compare the beck depression and anxiety values of the nulliparous and multipar pregnant women who undergo optional abortion below 12 weeks and to evaluate the effect of the parity on depression and anxiety.

DETAILED DESCRIPTION:
The beck depression and anxiety scale consists of questionnaire questions asked to the patient, and the value on 17 indicates advanced depression.

The BDI inventory has maximum of 63 and minimum of 0 scores:

(0-10): Are considered normal ups and downs (11-16): Mild mood disturbance (17-20): Borderline clinical depression (21-30): Moderate depression, (31-40): Severe depression, Over 40: Extreme depression. A persistent score of !17, requires psychiatric treatment

ELIGIBILITY:
Inclusion Criteria:

* healthy
* Women with a pregnancy less than 12 weeks
* no psychiatric disease or drug use

Exclusion Criteria:

* Those who have had a psychiatric diagnosis before,
* Women under the age of 18,
* Psychiatric drug users,
* Those who have experienced a major trauma or disease
* During the 3-month follow-up period, who developed complications during the procedure pregnant again
* Women with a pregnancy greater than 12 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Comparison of beck depression and anxiety values of nulliparous and multiparous pregnants who underwent optional abortion below 12 weeks and the effect of parity on depression and anxiety.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Beck Depression and Anxiety Scores in Multipar and Nulliparous Women who have gone under Dilatation and Curettage | 3 months
  to evaluate the effect of the parity on depression and anxiety.
  The BDI inventory has maximum of 63 and minimum of 0 scores:
  (0-10): Are considered normal ups and downs (11-16): Mild mood disturbance (17-20): Borderline clinical depression (21-30): Moderate depression, (31-40): Severe depression, Over 40: Extreme depression. A persistent score of !17, requires psychiatric treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Yalçın Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)